CLINICAL TRIAL: NCT06317025
Title: Design and Development of Multi-modal Intelligent Anesthesia Monitoring System
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SHOUFA2022-2Z-2039
Record Dates: First submitted 2024-02-21; First posted 2024-03-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia
Keywords: Anesthesia monitoring; Near infrared reflectance spectroscopy（NIRS）; electroencephalogram（EEG）; multimodal; Age dependent; Machine learning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anaesthetic patient: Monitoring depth of anaesthesia using PRST （P：pressure， T：tear，R：rate， S：sweat）score developed by Evans and bispectral index
  Interventions: Diagnostic Test: Multi-modal Intelligent Anesthesia Monitoring System

INTERVENTIONS:
Diagnostic Test: Multi-modal Intelligent Anesthesia Monitoring System — To evaluate the sensitivity and specificity of self-developed anesthesia monitoring systems in diagnosing the depth of anesthesia (too deep or too shallow)

SUMMARY:
This project integrates the characteristics of electroencephalo-graph（EEG）, cerebral oxygen, blood pressure, heart rate, etc., based on nonlinear theory and neural oscillation, large sample data and machine learning theory, to develop a multi-modal monitoring system suitable for domestic patients, taking into account changes in sedation, analgesia, cerebral hemodynamics and other factors, regardless of patient age and type of general anesthesia drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 0-65 years old
2. ASA: Level I-III
3. Patients undergoing non cardiac surgery under general anesthesia
4. Informed consent of the patient or legal representative

Exclusion Criteria:

1. Previous history of severe neurological disorders
2. History of mental illness and related medication use
3. Individuals who are unable to cooperate in completing cognitive function tests
4. Severe hearing or visual impairment
5. Preoperative delirium in patients
6. Individuals who have experienced severe adverse reactions such as cardiac arrest and cardiopulmonary resuscitation during surgery
7. Those who require neurosurgery, head and facial surgery
8. Individuals who are allergic to EEG and fNIRS electrodes

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing non-cardiac surgery under general anesthesia in Beijing Chaoyang Hospital, Capital Medical University
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
the depth of anesthesia (too deep or too shallow) | During general anesthesia
  PRST score system, combined with BIS index for comprehensive judgment

SECONDARY OUTCOMES:
EEG characteristics of loss of consciousness induced by different general anesthesia drugs | During general anesthesia
  Spectral Analysis，Connectivity Analysis，Brain Networks Analysis
Characteristics of perioperative neurovascular coupling | Perioperative
  EEG power and entropy indexes are extracted by moving window method as new time series, and a new time series consistent with NIRS is constructed. The entropy and power of different frequency bands after resampling were used as the indexes of neural activity, and ΔHbO and ΔHb were selected as the indexes of hemodynamic activity. The neurovascular coupling was evaluated by calculating the coherence of neural activity and hemodynamic activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No